CLINICAL TRIAL: NCT03050047
Title: A Multicenter Open-Label Single-Arm Multi-Cohort Phase I Study of Pharmacokinetics, Pharmacodynamics, Safety, and Immunogenicity of BCD-100 (JSC BIOCAD, Russia) in Patients With Advanced Solid Tumors
Brief Title: A Multicenter Open-Label Single-Arm Multi-Cohort Phase I Study of BCD-100 in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BCD-100-1
Record Dates: First submitted 2017-02-08; First posted 2017-02-10 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Melanoma; Lung Cancer; Renal Cell Carcinoma
MeSH Terms: conditions — Melanoma; Lung Neoplasms; Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- BCD-100 0.3 mg/kg (Experimental): Patients who receive BCD-100 in a dose of 0.3 mg/kg
  Interventions: Biological: BCD-100
- BCD-100 1 mg/kg (Experimental): Patients who receive BCD-100 in a dose of 1 mg/kg
  Interventions: Biological: BCD-100
- BCD-100 3 mg/kg (Experimental): Patients who receive BCD-100 in a dose of 3 mg/kg
  Interventions: Biological: BCD-100
- BCD-100 10 mg/kg (Experimental): Patients who receive BCD-100 in a dose of 10 mg/kg
  Interventions: Biological: BCD-100

INTERVENTIONS:
Biological: BCD-100 — Anti-PD1 monoclonal antibody

SUMMARY:
A Multicenter Open-Label Single-Arm Multi-Cohort Phase I Study of Pharmacokinetics, Pharmacodynamics, Safety, and Immunogenicity of BCD-100 (JSC BIOCAD, Russia) in Patients with Advanced Solid Tumors

ELIGIBILITY:
Inclusion Criteria:

1. Patient provides a written informed consent and is able to follow the requirements of the Protocol;
2. Age ≥ 18 years
3. Histologically confirmed cancer (well-documented test results; preferably, block specimens available):

   * unresectable (stage III/IV) or metastatic (stage IV) melanoma (the drug will be used as the first of subsequent therapy lines);
   * Locally advanced or metastatic NSCLC (squamous cell carcinoma/adenocarcinoma), progressive after at least the first-line therapy (the drug will be used as a second or subsequent therapy lines);
   * Metastatic clear cell renal carcinoma, progressive after at least the first-line therapy (the drug will be used as a second or subsequent therapy lines);

   In addition, by investigator's decision, patients with the following malignancies can also be enrolled in the study :
   * Pleural mesothelioma progressive after at least one therapy line (the drug will be used as a second or subsequent therapy lines);
   * Metastatic bladder cancer progressive after at least one therapy line (the drug will be used as a second or subsequent therapy lines);
   * Triple negative breast cancer (ER-, PR-, HER2-) progressive after at least the first-line therapy (the drug will be used as a second or subsequent therapy lines);
4. ECOG score of 0 to 2;
5. Measurable disease (at least one lesion) according to RECIST v. 1.1 ;
6. Resolved toxicity events from the previous therapy or adverse consequences of surgical interventions to ≤ grade 1 CTCAE v. 4.03, except for chronic/irreversible adverse events not affecting the safety of the study therapy (e.g. alopecia);
7. No severe pathology of organs or systems;
8. Life expectancy of at least 12 weeks from the screening;
9. Patients of childbearing potential enrolled in the study must agree to use reliable contraception methods throughout the study period, beginning 2 weeks before the inclusion in the study and up to 8 weeks after the last dose of BCD-100.

Exclusion Criteria:

1. Severe concomitant illnesses or life-threatening consequences (including pleural/pericardial/peritoneal effusion that requires medical intervention , pulmonary lymphangitis, or involvement of >50% renal parenchyma);
2. Brain metastases, progressive or associated with clinical symptoms (e.g. cerebral edema or spinal cord compression). Exclusions: metastases that do not progress and do not require steroids and/or anticonvulsants within at least 4 weeks before randomization ;
3. Severe cardiovascular disorders within 6 months before screening;
4. Autoimmune diseases;
5. Conditions requiring steroids or any other immunosuppressants;
6. Blood disorders: ANC ≤1,500/mm3; platelets ≤100,000/mm3; or Hb ≤90 g/L;
7. Renal function impairment: creatinine ≥1.5 × ULN;
8. Hepatic function impairment: bilirubin ≥1.5 × ULN; AST and ALT ≥2.5 × ULN (5 × ULN for patients with liver metastases), AlkPh ≥ 5 × ULN;
9. Prior anticancer treatment within 28 days before starting the study drug (surgery, radiation therapy , or chemotherapy);
10. Known history of more than 6 lines of systemic anticancer chemotherapy (including neoadjuvant and adjuvant CTs);
11. Prior treatment with anti-PD1/PDL1 agents or CTLA4 inhibitors;
12. Concurrent malignancy except for radically resected cervical carcinoma in situ or radically resected basal cell/squamous cell carcinoma;
13. Conditions limiting patient's ability to follow the Protocol requirements (dementia, neurological or psychiatric disorders, drug or alcohol abuse, etc.);
14. Simultaneous participation in any other clinical trial; participation in other clinical trials within 30 days before inclusion in the present study; previous participation in the present study.
15. Acute infections or active chronic infections;
16. Documented HIV infection;
17. Positive screening results for Hbs-antigen, hepatitis B core antibodies (anti-HBc Ab) and/or hepatitis C antibodies ;
18. Positive results of microprecipitation reaction together with positive TPHA assay results at the screening;
19. Body weight > 95 kg.
20. Intravenous administration of the drug is impossible;
21. Intravenous administration of contrast agents is impossible;
22. Hypersensitivity to any component of BCD-100.
23. Known history of hypersensitivity to monoclonal antibodies;
24. Pregnancy or breastfeeding;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-08-30 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
ORR (CR + PR) | 85 days
  Pilot efficacy assessment is not the primary objective of this study and will be conducted by surrogate endpoints describing the direct antitumor effect of the drug.
  • ORR (CR + PR) after 85 days of therapy with BCD-100.

CONTACTS AND LOCATIONS:
Locations (4):
- Russia (4):
  - "Russian Cancer Research Center named after N.N. Blokhin "of the Ministry of Health of the Russian Federation, Moscow
  - N.N.Petrov Oncology Research Center, Saint Petersburg
  - LLC BioEk, Saint Petersburg
  - State budgetary health care institution "St. Petersburg Clinical Scientific and Practical Center of Specialized Medical Assistance (Oncological)", Saint Petersburg